CLINICAL TRIAL: NCT00684489
Title: Renin-Guided Therapeutics in the Management of Untreated, Uncontrolled or Complicated Hypertension
Brief Title: Renin-Guided Therapeutics in the Management of Untreated, Uncontrolled, or Complicated Hypertension
Acronym: Renin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Brent M. Egan, MD, Medical University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11023; HR# 11023
Record Dates: First submitted 2008-02-25; First posted 2008-05-26 (Estimated); Last update posted 2008-05-26 (Estimated); Status verified 2008-05

CONDITIONS: Hypertension
Keywords: hypertension; renin-guided therapeutics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A; B (Active Comparator)
  Interventions: Drug: clinical hypertension specialist-no specific med. Any anti-hypertension meds.; Drug: renin guided therapeutics-no specific med. Any anti-hypertensive med.
- 2 (Active Comparator): Arm A is assignment to a clinical hypertension specialist Arm B is assigned renin-guided therapeutics
  Interventions: Drug: clinical hypertension specialist-no specific med. Any anti-hypertension meds.; Drug: renin guided therapeutics-no specific med. Any anti-hypertensive med.
- A is clinical hypertension specialist (Active Comparator): Arm A is assigned to a clinical hypertension specialist
  Interventions: Drug: clinical hypertension specialist-no specific med. Any anti-hypertension meds.
- Arm B is renin-guided therapeutics (Active Comparator): This group will be assigned to renin-guided therapeutics
  Interventions: Drug: renin guided therapeutics-no specific med. Any anti-hypertensive med.

INTERVENTIONS:
Drug: clinical hypertension specialist-no specific med. Any anti-hypertension meds. — assignment to a clinical hypertension specialist. Drugs used were hypertension medications were: chlorothiazide, hydrochlorothiazide, polythiazide indapamide, metolazone, bumetanide, furosemide, torsemide, amiloride, triamterene, eplerenone, spironolactone, atenolol, betaxolol, bisoprolol, metoprolol, nadolol, propranolol, timolol, acebutolol, penbutolol pindolol, carvedilol, labetalol, benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan, diltiazem, dilacor, ditiazem, verapamil, amlodipine, felodipine, isradipine, nicardipine, nifedipine, nisoldipine, doxazosin, prazosin, terazosin, clonidine, clonidine patch, methyldopa, reserpine, guanfacine, hydralazine, minoxidil.
  Arms: 2; A is clinical hypertension specialist; A; B
Drug: renin guided therapeutics-no specific med. Any anti-hypertensive med. — renin guided therapeutics-chlorothiazide, chlorthalidone, hydrochlorothiazide, polythiazide, indapamide, metolazone, bumetanide, furosemide, torsemide, amiloride, triamterene, eplerenone, spironolactone, atenolol, betaxolol, bisoprolol, metoprolol, nadolol, propranolol, timolol, acebutolol, penbutolol, pindolol, carvedilol, labetalol, benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan, diltiazem, dilacor, verapamil, amlodipine, felodipine, isradipine, nicardipine, nifedipine, nisoldipine, doxazosin, prazosin, terazosin, chlonidine, methyldopa, reserpine, guanfacine, hydralazine, minoxidil.
  Arms: 2; A; B; Arm B is renin-guided therapeutics

SUMMARY:
Plasma renin values determine whether volume or vasoconstrictor (renin) factors predominate in elevating blood pressure and are useful in selecting effective antihypertensive therapy.2,3

The researchers hypothesize that:

1. Plasma renin-guided therapeutics will improve systolic and diastolic blood pressure control in patients with untreated hypertension as well as in patients with treatment refractory or resistant hypertension that are managed by Clinical Hypertension Specialists.
2. Renin-guided therapeutics will reduce the number of medications required to maintain blood pressure control to <140/90 mmHg in hypertensive patients receiving 3 or more medications, while under the care of a Clinical Hypertension Specialist.
3. Renin-guided therapeutics selection will reduce the total cost of antihypertensive care provided by Clinical Hypertension Specialists.

DETAILED DESCRIPTION:
Hypertension affects ~25% of adults. The prevalence of hypertension and related complications is greater among the elderly, obese, and ethnic minorities. Unfortunately, hypertension control rates remain in the 25% range and are often significantly lower for the high-risk groups noted.1 Since the high-risk groups are growing more rapidly than the general population, the prevalence of hypertension and associated morbidity and mortality will probably increase sharply in the years ahead unless successful strategies are implemented for dramatically improving blood pressure control.

Direct measurements of plasma renin reflect the relative balance between volume (V) and vasoconstrictor (renin [R]) factors underlying the elevated blood pressure in patients with essential hypertension.2 While many antihypertensive medications have effects on both the volume (V) and vasoconstrictor (renin [R]) components of elevated blood pressure, one or the other usually predominates

ELIGIBILITY:
Inclusion Criteria:

* Age, 21 years of age and older
* Male or female (post-menopausal or effective method of birth control)
* BP and treatment criteria noted above
* Willingness to provide written, informed consent
* Ability to adhere to study protocol

Exclusion Criteria:

* Uncontrolled diabetes or hyperlipidemia requiring medication changes
* Any active disease process requiring new diagnostic and therapeutic plans
* Any life-threatening illness
* History of alcohol or drug abuse in past 5 years
* Mental illness or personality disorder that interfere with adherence to study protocol
* Serum creatinine >2.5 mg/dL unless documented stable for at least one year
* Dialysis for chronic renal failure, even if creatinine stable for at least one year
* Intolerance to two or more classes of antihypertensive medications
* Normal home BP (<140/90 mmHg at baseline), i.e., office only hypertension.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-09; Primary Completion 2005-03 (Actual); Study Completion 2005-09 (Actual)